CLINICAL TRIAL: NCT04885400
Title: iJobs - Testing the Feasibility and Acceptability of an Online Adaptation of the Jobs Program: an Open-label Pilot Study
Brief Title: Feasibility and Acceptability of the Online JOBS Program
Acronym: iJobs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: iJobs
Record Dates: First submitted 2021-04-28; First posted 2021-05-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2021-04

CONDITIONS: Unemployment

STUDY DESIGN:
Intervention Model Description: Open-label pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iJobs (Experimental): All the participants will be included in the program.
  Interventions: Behavioral: iJobs

INTERVENTIONS:
Behavioral: iJobs — During the program, the participants will learn and exercise successful job search strategies. The web-based adaptation of the Jobs program will allow self-administration. After each session, they will receive written feedback from trainers on the platform.

SUMMARY:
The aim of this study is to test the feasibility and acceptability of a web-based adaptation of the Jobs program (developed by Curran et al., 1999).

DETAILED DESCRIPTION:
The current study is an open trial that will test the feasibility and acceptability of a web-based adaptation of the Jobs program (further be referred to as iJobs). We will use a repeated measures design: one group and three measurements (baseline, post-intervention, 3 months follow-up). iJobs consists of five sessions spread over a two-week period. The participants will learn and exercise successful job search strategies (e.g. finding job openings, creating an attractive resume, demonstrating effective interviews).

ELIGIBILITY:
Inclusion Criteria:

* Unemployed and looking for a job
* Work as volunteers and looking for a paid job
* Have a PC or laptop and basic digital competencies

Exclusion Criteria:

* They don't have internet access and are not available during the two weeks of the program
* Suffer from a chronic disease that implies special conditions for taking part in the activities
* Severe clinical depression symptoms (Cut-off=15 at PHQ9)*
* Severe clinical anxiety symptoms (Cut-off=15 at GAD7)*

(*) will be included if they receive mental health treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Job search behavior effort | Change from baseline to follow-up (3 months).
  Job search behavior effort: Job Search Behavior Scale (Blau, 1994) was designed to measure participants' involvement in job search activities, in terms of frequency and intensity. The minimum score is 16 and the maximum is 80. A higher score means a better outcome (increased job search behavior effort).
Satisfaction with the intervention | Post-intervention (2 weeks).
  Satisfaction with the intervention will be measured using 22 items. We will use 6 items aiming at the program's content retrieved from a questionnaire used for measuring the alliance between trainers and trainees in a face-to-face JOBS intervention. The minimum score is 6 and the highest is 42. A higher score means a better outcome (increased satisfaction with the intervention). Also, we will use 16 items retrieved from a scale previously used for measuring the satisfaction with an online intervention delivered on the same platform as we will use for our program. Nine of the items are measured on a Likert scale. The minimum score is 7 and the maximum is 42. A higher score means greater satisfaction. 7 items are open-ended questions and imply qualitative analysis.
System usability | Post-intervention (2 weeks).
  We will use a 10 item questionnaire (Bangor et al., 2009) designed to measure participants' satisfaction with e-cbt, the online platform used for the program delivery. The total score of System Usability Scale is 0 and the highest one is 100. A higher score means a better outcome.
Treatment adherence | Post-intervention only (2 weeks).
  The number of completed assignments; Quality of completed assignment (qualitative rating of the degree of completeness and depth of the answer for each assignment, conducted by two independent experts based on apriori established coding grids).

SECONDARY OUTCOMES:
Job-Search Self-Efficacy | Change from baseline to post-intervention (2 weeks).
  Job Search Self-Efficacy Scale was designed to measure participants' perception of their ability to gain employment. We will use the 20 item version of the scale developed by Saks et al., 2015. The minimum score is 20 and the maximum is 100. A higher score means a better outcome (increased job search self-efficacy).
Self-esteem | Change from baseline to post-intervention (2 weeks).
  Rosenberg's Self Esteem Scale is a self-esteem measure widely used in social science research. It is a ten-item Likert-type scale with items answered on a four-point scale-from strongly disagree to strongly agree. The scale measures global self-worth by measuring both positive and negative feelings about the self. The minimum score of Rosenberg's Self Esteem Scale is 10 and the highest one is 40. A higher score means a better outcome.
Inoculation against setbacks | Change from baseline to post-intervention (2 weeks).
  We will use 2 items retrieved from previous studies (Vuori & Vinokur, 2005) aiming to measure the effectiveness of JOBS intervention in terms of participant's ability to deal with setbacks. The minimum score is 2 and the maximum is 10. A higher score means a better outcome (presence of inoculation against setbacks).
Future Career Anxiety | Change from baseline to post-intervention (2 weeks).
  We will measure participant's anxiety regarding their future career in the context of the COVID-19 outbreak with the Future Career Anxiety Scale developed by Tsai et al., 2017 (Mahmud et al., 2020). The minimum score is 5 and the maximum is 25. A higher score means a worse outcome (increased anxiety).
Patient Health Questionnaire-9 (PHQ9) | Change from baseline to post-intervention (2 weeks).
  Patient Health Questionnaire-9 was designed to measure participants' severity of depression using DSM IV criteria. The minimum score of Patient Health Questionnaire-9 is 0 and the highest one is 27. A higher score means a worse outcome (more severe symptoms of depression).
Generalised Anxiety Disorder Assessment (GAD7) | Change from baseline to post-intervention (2 weeks).
  Generalised Anxiety Disorder Assessment is a self-administered 7 item instrument that uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. The minimum score of Generalised Anxiety Disorder Assessment is 0 and the highest one is 21. A higher score means a worse outcome (a higher level of anxiety).
Employment status | Follow-up (3 months).
  Self-reported employment status (phone screening).
Job Quality | Follow-up (3 months).
  For those who found employment - phone screening.

OTHER OUTCOMES:
Physical health | Baseline only (factors to be controlled for).
  We will use a short-version of the Physical Health Complaints Scale (Ware, 1999) to measure participants' perception of their health. The minimum score is 4 and the highest is 20. A higher score means a worse outcome (worse physical health).
Financial strain | Baseline only (factors to be controlled for).
  We will use a single item from Vuori & Vinokur, 2005 to assess participants' financial strain, respectively: 'What is the financial situation of your family/household in your opinion?'. The minimum score is 1 while the maximum is 5. A higher score means a high level of financial strain.
Sociodemographic information | Baseline only
  Age, gender, background, educational level, average monthly income, unemployment period, work experience, and targeted professional field.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Rusu, Principal Investigator — West University of Timisoara
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Bangor, A.,Kortum, P. & Miller, J. (2009). Determining what individual SUS scores mean: adding an adjective rating scale. Journal of Usability Studies, 4(3), 114-123.
- [Background] Blau, G. (1994). Testing a Two-Dimensional Measure of Job Search Behavior. Organizational Behavior and Human Decision Processes, 59(2), 288-312. https://doi.org/10.1006/obhd.1994.1061
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Mahmud MS, Talukder MU, Rahman SM. Does 'Fear of COVID-19' trigger future career anxiety? An empirical investigation considering depression from COVID-19 as a mediator. Int J Soc Psychiatry. 2021 Feb;67(1):35-45. doi: 10.1177/0020764020935488. Epub 2020 Jul 2. PMID 32615833
- [Background] Rosenberg, M. (1979). Conceiving the Self. New York: Basic Books.
- [Background] Saks, A.M., Zikic, J. & Koen, J. (2015). Job search self-efficacy: Reconceptualizing the construct and its measurement. Journal of Vocational Behavior, 86, 104-114. https://doi.org/10.1016/j.jvb.2014.11.007
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ware JE Jr, Keller SD, Hatoum HT, Kong SX. The SF-36 Arthritis-Specific Health Index (ASHI): I. Development and cross-validation of scoring algorithms. Med Care. 1999 May;37(5 Suppl):MS40-50. doi: 10.1097/00005650-199905001-00004. PMID 10335742
- [Background] Vuori, J. & Vinokur, A.D. (2005). Job-search preparedness as a mediator of the effects of the Tyohon Job Search Intervention on re-employment and mental health. Journal of Organizational Behavior, 26, 275-291. DOI: 10.1002/job.308